CLINICAL TRIAL: NCT03769155
Title: Pilot Integrated Biomarker Study of VX15/2503 in Combination With Ipilimumab or Nivolumab in Patients With Resectable Metastatic Melanoma
Brief Title: VX15/2503 With or Without Ipilimumab and/or Nivolumab in Patients With Resectable Stage IIIB-D Melanoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Vaccinex Inc. (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Lowe, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00104273; NCI-2018-01229 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4400-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8
MeSH Terms: interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; pepinemab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- A (VX15/2503, nivolumab, surgery) (Experimental): Participants receive VX15/2503 (pepinemab) IV over 60 minutes and nivolumab IV over 30 minutes on days 1 and 21 and undergo surgery between days 35-49.
  Interventions: Biological: Nivolumab; Biological: VX15/2503; Procedure: Surgery
- B (VX15/2503, ipilimumab, surgery) (Experimental): Participants receive VX15/2503 (pepinemab) IV over 60 minutes and ipilimumab IV over 30 minutes on days 1 and 21 and undergo surgery between days 35-49.
  Interventions: Biological: Ipilimumab; Biological: VX15/2503; Procedure: Surgery
- C (VX15/2503, nivolumab, ipilimumab, surgery) (Experimental): Participants receive VX15/2503 (pepinemab) IV over 60 minutes, nivolumab IV over 30 minutes, and ipilimumab IV over 30 minutes on days 1 and 21 and undergo between days 35-49.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Biological: VX15/2503; Procedure: Surgery
- D (nivolumab, surgery) (Experimental): Participants receive nivolumab IV over 30 minutes on days 1 and 21 and undergo between days 35-49.
  Interventions: Biological: Nivolumab; Procedure: Surgery
- E (surgery) (Active Comparator): Participants undergo surgery.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: B (VX15/2503, ipilimumab, surgery); C (VX15/2503, nivolumab, ipilimumab, surgery)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: A (VX15/2503, nivolumab, surgery); C (VX15/2503, nivolumab, ipilimumab, surgery); D (nivolumab, surgery)
Biological: VX15/2503 — Given IV
  Other Names: moAb VX15/2503; Pepinemab
  Arms: A (VX15/2503, nivolumab, surgery); B (VX15/2503, ipilimumab, surgery); C (VX15/2503, nivolumab, ipilimumab, surgery)
Procedure: Surgery — Undergo therapeutic conventional surgery

SUMMARY:
This pilot phase I trial studies how well VX15/2503 (pepinemab) with or without ipilimumab and/or nivolumab work in treating participants with stage IIIB-D melanoma that can be removed by surgery. Monoclonal antibodies, such as VX15/2503, ipilimumab, and nivolumab may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the effect of VX15/2503 (pepinemab) in combination with immune checkpoint inhibitors on T cell infiltrate into the tumor microenvironment in involved and uninvolved lymph nodes and peripheral blood.

SECONDARY OBJECTIVES:

I. Evaluate the effect of VX15/2503 in combination with immune checkpoint inhibitors on the immune profile of involved and uninvolved lymph nodes and peripheral blood.

II. Assess safety and tolerability of profile and tolerability of single agent VX15/2503 to the combination of VX15/2503 and immune checkpoint inhibitors in patients with resectable metastatic melanoma.

III. Document pathologic response rates of single agent VX15/2503 and combination VX15/2503 and immune checkpoint inhibitors in patients with resectable melanoma.

IV. Compare pathologic response to radiographic response using Response Evaluation Criteria in Solid Tumors (RECIST) criteria in patients receiving single agent VX15/2503 and combination VX15/2503 and immune checkpoint inhibitors in patients with resectable melanoma.

OUTLINE: Participants are assigned to 1 of 5 arms.

ARM I: Participants receive VX15/2503 intravenously (IV) over 60 minutes and nivolumab IV over 30 minutes on days 1 and 21 and undergo surgery between days 35-49.

ARM II: Participants receive VX15/2503 IV over 60 minutes and ipilimumab IV over 30 minutes on days 1 and 21 and undergo surgery between days 35-49.

ARM III: Participants receive VX15/2503 IV over 60 minutes, nivolumab IV over 30 minutes, and ipilimumab IV over 30 minutes on days 1 and 21 and undergo between days 35-49.

ARM IV: Participants nivolumab IV over 30 minutes on days 1 and 21 and undergo between days 35-49.

ARM V: Participants undergo surgery.

After completion of study treatment, participants are followed up at 90 days, every 12 weeks for 2 years, every 6 months for 3 years, then annually up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB, IIIC, IIID histologically-proven melanoma.

  * Cancer confirmed to be surgically resectable, with surgery evaluation with planned prior to resection.
  * No prior immunotherapy with cytotoxic T-lymphocyte associated protein-4 (CTLA-4), anti programmed cell death-1 (PD-1) or VX15/2503. Prior interferon (at least 1 year prior to consent) will be allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Absolute neutrophil count ≥ 1,500 cells/µL.
* Platelets ≥ 100,000/µL.
* Hemoglobin ≥ 9.0g/dL (may receive packed red blood cells [PRBC] transfusion).
* Total bilirubin ≤ 1.5 x the upper limit of normal (ULN).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN.
* Albumin ≥ 3.0 g/dL.
* Serum creatinine ≤ 1.5 x ULN OR calculated creatinine clearance of ≥ 50 mL/min using Cockcroft-Gault formula.
* International normalized ration (INR) ≤ 1.5. Anticoagulation is allowed only with low molecular weight heparin (LMWH). Patient receiving LMW heparin on stable therapeutic dose for more than 2 weeks or with factor Xa level < 1.1 U/mL are allowed on the trial.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Ability to understand and willingness to sign a written informed consent document.
* Female subjects of childbearing potential must agree to use adequate contraception (at least one highly effective method and one additional method of birth control at the same time or complete abstinence) prior to study entry, for the duration of study treatment and 5 months after last dose of study treatment.
* Male subjects must agree to use adequate contraception (at least one highly effective method and one additional method of birth control at the same time or complete abstinence) prior to study entry, for the duration of study treatment and 7 months after last dose of study treatment.
* Female subjects of childbearing age must have a negative serum pregnancy test at study entry.

Exclusion Criteria:

* Determined not to be a surgical candidate due to medical co-morbidities.
* Treatment with chronic immunosuppressants (e.g., cyclosporine following transplantation).
* Prior organ allograft or allogeneic bone marrow transplantation.
* Subjects with active or history of immune mediated pneumonitis, colitis, hepatitis, endocrinopathy, nephritis, or skin reactions as these patients may be at increased risk for developing immune therapy-induced exacerbation or recurrence of their immune mediated disease, potentially delaying surgery.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Women who are pregnant or lactating.
* Uncontrolled intercurrent illness including, but not limited to, human immunodeficiency virus (HIV)-positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure (NYHA class III or IV), unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Other medications, or severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Clinical evidence of bleeding diathesis or coagulopathy.
* Patients with prior malignancies, including pelvic cancer, are eligible if they have been disease free for > 5 years. Patients with prior non-melanoma skin cancers and in situ carcinomas are eligible provided there was complete removal.
* Active bacterial or fungal infections requiring systemic treatment within 7 days of treatment.
* Use of other investigational drugs (drugs not marked for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration.
* History of severe hypersensitivity reactions to other monoclonal antibodies.
* Non-oncology vaccines within 28 days prior to or after any dose of ipilimumab.
* Prisoners and subjects who are compulsory detained.
* Patients with rapidly progressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2032-12-15 (Estimated)

PRIMARY OUTCOMES:
Biomarker parameter analysis: extent of cluster of differentiation 8 (CD8)+ T cell infiltration between experimental groups following treatment | Up to 10 years after study start
  The two-sample t-test will be used to compare the change in CD8+ T cell infiltration after treatment between each experimental group (Cohort A, B, C, and D) and the control group (cohort E), respectively.

SECONDARY OUTCOMES:
Incidence of adverse events assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 8 weeks after surgery
  Descriptive statistics for worst grade of each laboratory parameter by the NCI CTCAE scale version 4.0 at baseline and follow-up will be presented.
Response rate | Up to 10 years after study start
  For participants to be considered evaluable for efficacy, they must have completed the treatment and have a baseline tumor assessment. Response rate will be calculated as proportion (responders/total participants).
Overall survival (OS) | Assessed up to 10 years after study start
  For overall survival, death from any cause will be defined as the event.
Progression-free survival (PFS) | Assessed up to 10 years after study start
  Progression or death from any cause will be defined as the event.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lowe, MD, MA, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03769155/ICF_000.pdf